CLINICAL TRIAL: NCT05228119
Title: A Single-Arm, Open-Label, Exploratory Study to Evaluate Safety and Efficacy of Oncolytic Virus Injection (RT-01) in Combination With PD-1 Inhibitor (Nivolumab) in Patients With Advanced Solid Tumors
Brief Title: A Study of Oncolytic Virus Injection (RT-01) in Combination With PD-1 Inhibitor in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LWY21076CXY
Record Dates: First submitted 2022-01-03; First posted 2022-02-08 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Advanced Solid Tumor
Keywords: RT-01; Oncolytic Virus; PD-1 Inhibitor; immunotherapy; immune Checkpoint Inhibitors; Intravenous Injection; Intratumoral injection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oncolytic Virus Injection(RT-01) (Experimental): RT-01 will be administered either intravenously or with a combination of intravenously and intratumorally on day 1.
  Nivolumab will be administered intravenously every 3 weeks starting on day 5.
  Interventions: Biological: Oncolytic Virus Injection(RT-01)

INTERVENTIONS:
Biological: Oncolytic Virus Injection(RT-01) — Intravenous injection with or without intratumoral injection of a single dose of RT-01 and intravenous infusion of Nivolumab

SUMMARY:
This is a single-arm, open-label, exploratory study to evaluate safety and efficacy of oncolytic virus injection(RT-01) in combination with PD-1 inhibitor (Nivolumab) in patients with advanced solid tumors.

The purpose of this study is to evaluate the safety and tolerability, antitumor activity, The immunoreactivity, The immunogenicity, pharmacokinetics and virus shedding of RT-01 in combination with PD-1 inhibitor.

DETAILED DESCRIPTION:
This is an investigator initiated , single-arm, open-label study of RT-01 as a single agent given via Intravenous injection（IV）with or without Intratumoral injection（IT） in combination with IV Nivolumab in patients with advanced solid tumors.

This study is planned to enroll 40-50 patients with advanced solid tumors. RT-01 will be administered as a single dose on day 1, Nivolumab will be administered intravenously every 3 weeks starting on day 5.

The purpose of this study is to assess the safety and tolerability, antitumor activity, The immunoreactivity, The immunogenicity, pharmacokinetics and virus shedding of RT-01 in combination with PD-1 Inhibitor (Nivolumab).

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥ 18 years;
* Subjects must have histologically or cytologically confirmed diagnosis of advanced solid tumor(s) who have failed in standard therapy (disease progression or intolerance) and no effective treatment, or have no standard therapy, or have failed to obtain standard treatment due to objective conditions ;
* Subjects have At least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1) (non-nodal lesions with longest diameter ≥ 10 mm, or nodal lesions with short diameter ≥ 15 mm);
* ECOG score of 0 ~ 2;
* Adequate bone marrow, hepatic and renal and coagulation function;
* Women of childbearing age who have a negative pregnancy test within 7 days before treatment. Female patients of childbearing age, and male patients with partners of childbearing age must agree to use at least one medically recognized contraceptive method during study treatment and within at least 6 months after the last dose of investigational drug;
* Voluntarily participated in this study, signed the informed

Exclusion Criteria:

* Subjects with known brain metastasis and/or clinically history tumor brain of metastasis；
* Subjects who have received anti-tumor therapy such as chemotherapy, radiotherapy, biological therapy, endocrine therapy, targeted therapy, immunotherapy, etc within 2 weeks before RT-01 administration；
* Subjects who have participate in another interventional study within 4 weeks before RT-01 administration；
* Subjects who have had major surgery within 4 weeks before RT-01 administration；
* Patients in any condition requiring systemic treatment with corticosteroids (prednisone > 10 mg/day or equivalent of the similar drug) or other immunosuppressive agents within 14 days before RT-01 administration, but currently or previously treated with any of the following steroid regimens, were included: Topical, ophthalmic, intra-articular, intranasal, or inhaled corticosteroids with minimal systemic absorption; Prophylactic short-term use of corticosteroids；
* Subjects who have participate in another oncolytic virus study within 8 weeks before RT-01 administration；
* Subjects received live vaccines within 7 days before RT-01 administration；
* Subjects received Antiviral drugs within 2 weeks, long-acting interferon within 4 weeks before RT-01 administration；
* Subjects with adverse reactions caused by previous anti-tumor treatment not recovered to (CTCAE 5.0) grade 1 (except alopecia);
* Subjects who have uncontrolled active infection;
* Subjects with known positive history of human immunodeficiency virus (HIV) test or known acquired immunodeficiency syndrome (AIDS);
* Subjects who have active hepatitis;
* Subjects who have serious cardiovascular system disorders history;
* Subjects with active autoimmune diseases or history of autoimmune diseases that may relapse;
* Subjects having any serious uncontrolled disease or in other conditions that would preclude them from receiving study treatment and are considered unsuitable for this study in the opinion of the investigator;
* Subjects in other conditions that are considered unsuitable for this study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-01-04 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 6 months
  Graded according to the NCI CTCAE version 5.0.
Objective response rate | Up to 2 years
  Assess the proportion of patients who achieved complete or partial response
Disease control rate | Up to 2 years
  Assess the proportion of patients who achieved complete or partial or stable response
The changes from baseline of lymphocyte counts | Up to 28 days
  The changes from baseline of Peripheral blood lymphocyte subtypes counts
The concentration of antiviral antibody. | Up to 22 Weeks
  The concentration of antiviral antibody of RT-01 in blood
The rate of subjects with viral shedding of RT-01 | Up to 22 Weeks
  The rate of subjects with viral RNA in the secretion
The Tmax of Viral RNA in blood | Up to 22 Weeks
  Time to peak viral RNA concentration
The Cmax of Viral RNA in blood | Up to 22 Weeks
  The peak viral RNA concentration

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No